CLINICAL TRIAL: NCT07234890
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Exploratory Study to Evaluate the Neuroprotective Effects of AV-001 on Hemodialysis-induced Brain Injury Via Cerebrovascular Stabilization in Chronic Hemodialysis Patients
Brief Title: Study to Evaluate the Effects of AV-001 on HD-induced Brain Injury.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute (Other)
Responsible Party: Principal Investigator, Chris McIntyre, MBBS DM, London Health Sciences Centre Research Institute
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 15976
Record Dates: First submitted 2025-09-25; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis

STUDY DESIGN:
Intervention Model Description: Double-Blind, Placebo Controlled, Exploratory Group 1 (N-20) Placebo Group 2 (N-20) AV-001 Low dose Group 3 (N-20) Av-001 High dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Placebo (Experimental): Participants randomized into one group 1placebo. Placebo will be administered 60 minutes prior to hemodialysis initiation, 3 x over a one-week treatment period.
  Interventions: Drug: AV-001 or Placebo Injection
- Group 2: AV-001 low dose (12.5μg/kg) (Experimental): Participants randomized into group 2 will receive AV-001 low dose. AV-001 low dose will be administered 60 minutes prior to hemodialysis initiation, 3 x over a one-week treatment period.
  Interventions: Drug: AV-001 or Placebo Injection
- Group 3: AV-001 High Dose (25μg/kg) (Experimental): Participants randomized into group 3 will receive AV-001 high dose. AV-001 high dose will be administered 60 minutes prior to hemodialysis initiation, 3 x over a one-week treatment period.
  Interventions: Drug: AV-001 or Placebo Injection

INTERVENTIONS:
Drug: AV-001 or Placebo Injection — AV-001 or Placebo administered via IV bolus injection.

SUMMARY:
Cognitive decline is increasingly recognized among patients receiving maintenance hemodialysis (HD). This can include trouble remembering, slower thinking or mentally feeling foggy.

This research is being done to determine if a new medication (AV-001) can protect the brain from injury caused by hemodialysis by strengthening blood vessels in the brain and reducing inflammation.

If successful, this research could lead to better protection for the brains of people undergoing regular dialysis, potentially reducing the risk of cognitive decline and stroke.

DETAILED DESCRIPTION:
Hemodialysis provides life-sustaining treatment for many chronic kidney disease patients around the world. Moderate to severe cognitive impairment is very common in HD patients with up to 70% being affected who are ≥ 55 years of age and ~ 10% in those between 21-39 years of age. Significant cognitive impairment is evident within 6 months of starting HD.

This study is a phase 2 exploratory study in patients receiving hemodialysis treatments. Investigators will recruit 60 patients from the renal program at the London Health Sciences Centre.

Study participants will receive AV-001 (low or high dose) or placebo 60 minutes prior to HD initiation at 3 HD treatment sessions within 1 week (Monday, Wednesday and Friday)

Study participants will also undergo:

* Vital sign collection (blood pressure and heart rate)
* Blood collection
* Cognitive assessments
* Vascular ultrasound
* MRI

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Male and non-pregnant female patients (>18 years old)
* HD for ≥ 3 months
* Thrice weekly HD schedule

Exclusion Criteria:

* HD <90 days
* Contraindication to MRI
* Established severe cognitive impairment (Montreal Cognitive Assessment test (MoCA) <18 or formal diagnosis of dementia)
* Previous clinical stroke
* Pregnancy, breastfeeding, or intending pregnancy
* Intradialytic hypotension event (defined as: drop in SBP ≥40mmHg + symptoms + intervention) in previous month as evidenced by HD record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of AV-001 (high dose, low dose) on structural brain injury associated with HD, using MRI as compared to placebo controls. | Before and after dialysis on study visit day 3.
  We will assess brain structure using MRI, allowing accurate detailed study of brain WM structural integrity.

SECONDARY OUTCOMES:
Evaluate circulating biomarkers of vascular injury (S-100β ) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  Blood Samples (S-100β) will be collected Pre-HD, Peak-HD and Post HD for analysis.
Evaluate circulatory biomarkers of vascular injury (transthyretin) | Study Visit Day 1 to Study Visit Day 3 (over a 1-week period)
  Blood samples (transthyretin) will be collected Pre-HD, Peak HD and Post HD for analysis.
Evaluate circulatory biomarkers of vascular injury (TNF-a) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  Blood Samples (TNF-a) will be collected Pre-HD, Peak-HD and Post HD for analysis
Evaluate circulatory biomarkers of vascular injury (IL-6) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  Blood samples (IL-6) will be collected Pre-HD, Peak-HD and Post HD for analysis
Evaluate circulatory biomarkers of vascular injury (serum lipopolysaccharide) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  Blood Samples (serum lipopolysaccharide) will be collected Pre-HD, Peak-HD and Post HD for analysis
Evaluate circulatory biomarkers of vascular injury (complete blood count) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  Blood Samples (complete blood count) will be collected Pre-HD, Peak-HD and Post HD for analysis.
Evaluate circulatory biomarkers of vascular injury (urea) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  Blood Samples (urea) will be collected Pre-HD, Peak-HD and Post HD for analysis.
Evaluate circulatory biomarkers of vascular injury (electrolytes) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  Blood Samples (electrolytes) will be collected Pre-HD, Peak-HD and Post HD for analysis.
Evaluate circulating biomarkers of vascular injury (dialysate composition) | Study Visit Day 1 to Study Visit Day 3 (over a 1-week period)
  Dialysate composition (sodium, potassium, calcium, magnesium, glucose) will be collected Pre-HD, Peak-HD and Post HD for analysis.
Evaluate circulatory biomarkers of vascular injury (Clot) | Study visit Day 1 to Study Visit Day 3 (over a 1-week period)
  Blood Samples (clot-troponin T and C-reactive protein) will be collected Pre-HD, Peak-HD and Post HD for analysis.
Evaluate circulatory biomarkers of vascular injury (AV-001 specific biomarkers) | Study Visit Day 1 to Study Visit Day 3. (over a 1-week period)
  AV-001 specific circulatory biomarkers (soluble Tie2, CXCL10, MCP-1, Angiopoietin-1, Angiopoietin-2) will be collected Pre-HD, Peak-HD and Post HD for analysis.
Evaluate variations in cognitive assessment performance scores using Montreal Cognitive Assessment (MoCA) | Study Visit Day 1 to Study Visit Day 3 (1 week)
  The Montreal Cognitive Assessment (MoCA) is validated and highly sensitive for the detection of mild cognitive impairment and measures short term memory; visuospatial abilities; executive function; attention; concentration and working memory; language; and orientation to time and place.
Evaluate variations in cognitive assessment performance scores using Trailsmaking Test A | Study Visit Day 1 to Study Visit Day 3 (1 week)
  The Trailsmaking 'A' Test is sensitive to various neurological impairments and provide information on visual search, scanning, speed of processing, mental flexibility and executive functions.
  The patient is asked to connect numbers 1 through 25 as quickly as possible.
Trailsmaking B (TMTB) | Study Visit Day 1 to Study Visit Day 3 (1 week)
  The Trailsmaking 'B' Test is sensitive to various neurological impairments and provide information on visual search, scanning, speed of processing, mental flexibility and executive functions. Patients are asked to alternate numbers and letters which requires thinking flexibility and mental shifting.
Evaluate variations in cognitive performance scores using Creyos | Study Visit Day 1 to Study Visit Day 3 (1 week)
  Creyos encompass assessments of short-term memory, reasoning, attention and verbal ability. Creyos is an online platform and will be completed on a study designated tablet.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD/PhD, Principal Investigator — London Health Science Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided